CLINICAL TRIAL: NCT00352950
Title: An Open-Label Clinical Trial Evaluating the Safety and Pharmacodynamics of Sirolimus and Panitumumab in Subjects With Advanced Non-Small Cell Lung Cancer
Brief Title: Safety Evaluation of Panitumumab and Sirolimus in Advanced Non-Small Cell Lung Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20040145
Record Dates: First submitted 2006-04-06; First posted 2006-07-17 (Estimated); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Oncology; Non-Small Cell Lung Cancer
Keywords: NSCLC, Lung cancer; Panitumumab; Sirolimus; mTOR; Monoclonal antibody
MeSH Terms: conditions — Neoplasms; Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

INTERVENTIONS:
Drug: AMG 954/Panitumumab

SUMMARY:
To determine the dose and schedule of sirolimus when given in combination with panitumumab in adult subjects with Stage IIIB/IV NSCLC

ELIGIBILITY:
Inclusion Criteria:

* Histologically- or cytologically-confirmed diagnosis of stage IIIB or IV Non-Small Cell Lung Cancer
* Received only one prior treatment (not including radiation)
* Measurable disease per Response Evaluation Criteria in Solid Tumors Group (RECIST) guidelines
* Life expectancy of ≥ 4 months
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate hematologic, renal and hepatic function
* Serum-fasting cholesterol ≤ 300 mg/dL Serum-fasting triglycerides ≤ 2.5 X ULN Exclusion Criteria:
* Brain metastases requiring treatment
* History of interstitial pneumonitis or pulmonary fibrosis or evidence of interstitial pneumonitis or pulmonary fibrosis on baseline
* Systemic chemotherapy, radiotherapy, hormonal therapy or immunotherapy within 30 days before enrollment
* Prior epidermal growth factor receptor targeting agents with the exception of the small molecule EGFr tyrosine kinase inhibitors
* Prior anti-tumor therapies including prior experimental agents or approved anti-tumor small molecules and biologics of short serum half-life (less than 1 week) within 30 days before enrollment, or prior experimental or approved proteins/antibodies with longer serum half-life within 6 weeks before enrollment
* Prior therapy with sirolimus, sirolimus analogs
* Immunosuppressive agents within 28 days before enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-03; Study Completion 2008-02

PRIMARY OUTCOMES:
safety within the first 3 weeks

SECONDARY OUTCOMES:
pharmacodynamic analysis of mTOR

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com